CLINICAL TRIAL: NCT04653350
Title: Effects of High Intensity Multi-Modal Exercise Training on Bone Density and Functional Performance in Postmenopausal Women
Brief Title: High Intensity Multi-Modal Exercise Training in Postmenopausal Women
Acronym: HIT-MMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Huma Riaz, Associate Professor, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Huma Riaz
Record Dates: First submitted 2020-11-26; First posted 2020-12-04 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Postmenopausal Osteoporosis; Postmenopausal Osteopenia
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This will be a Single factor, Pretest-Postest Control group Design with parallel assignment of patients into two groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Females participating in a clinical trial will be kept blind with respect to their allocated exercise group. The assessor doing reporting for the DEXA scan will also be kept blind about the patient group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIT-MMEX Group (Experimental): In this group Supervised High intensity Progressive Resistance Training, High intensity weightbearing/Impact exercises and High challenging Balance Training will be given. 2 times/week for 40-50minutes session progressively over the duration of 8 months.
  Interventions: Other: High Intensity Exercises
- Control Group (Active Comparator): In this Group Supervised general fitness exercises including general body stretches, treadmill walking, mild to moderate intensity progressive resistance training & balance exercises will be given. 2 times/week for 40-50minutes session progressively over the duration of 8 months.
  Interventions: Other: General Exercises

INTERVENTIONS:
Other: High Intensity Exercises — Supervised High intensity Progressive Resistance Training, High intensity weightbearing/Impact exercises and High challenging Balance Training will be given. 2 times/week for 40-50minutes session progressively over the duration of 8 months.
  Arms: HIT-MMEX Group
Other: General Exercises — Supervised general fitness exercises including general body stretches, treadmill walking, mild to moderate intensity progressive resistance training & balance exercises will be given. 2 times/week for 40-50minutes session progressively over the duration of 8 months
  Arms: Control Group

SUMMARY:
in Pakistan 9.9 million people are osteoporotic and 7.2 million amongst them are women. Globally after every 3 seconds there is occurrence of fragility fracture.In Pakistan females carries different risk factors based on distinct culture, environment, diet and lifestyle. So there is dire need to conduct more high quality clinical trials at National level in order to establish strong evidence in favor of low cost but highly effective exercise protocols for such a significant public health issue.

DETAILED DESCRIPTION:
In postmenopausal age, women bones get weak and easily fracture after 50years. In Pakistan every other female is silently suffering from this disease leading to bone, joint pain and disability. This project is innovatively designed first time in Pakistan to target weak bones of women with high intensity, progressive exercise training. The objectives of this study are to determine the effects of a high intensity multi-modal exercise training on bone mineral density and functional performance in postmenopausal women.

After initial screening based on history, subjective fracture risk calculations and subjective osteoporosis screening. Females fulfilling criteria and willing to participate in exercise trial will be recruited in the study. At baseline, DEXA scan will be done for Femoral and lumbar bone density. All performance based testing for functional performance outcome measures would be done at baseline, after 3 months & after 6 months. Patient will be called twice a week for 8months and DEXA will be repeated after 8months of training. It is hypothesized that supervised exercise training will improve bone mineral density and functional performance in postmenopausal women with low bone mass.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Women, at least 3 years since last mensuration.
* Age: 45-70years
* Body mass index (BMI) <30kg/m2
* Community ambulant without walking aid
* Good general health
* Willing for exercise therapy

Exclusion Criteria:

* History of fragility fracture in addition to BMD T-score of -2.5 or less
* MMSE < 20
* Taking Hormone replacement therapy or steroids from last 1 year.
* Had participated in regular exercise for last 1 year
* Systemic illness: hyperthyroidism, hyperparathyroidism, Diabetes Mellitus, renal failure, any malignancy, extensive radiation exposure
* Any orthopedic injury/disorder hindering performance of exercise.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Femoral Neck BMD (FN BMD) | 8 Months
  Change from Baseline in Femoral Neck Bone Mineral Density measured by DEXA scan
Lumbar Spine BMD (LS BMD) | 8 Months
  Change from Baseline in Lumbar Spine Bone Mineral Density measured by DEXA scan

SECONDARY OUTCOMES:
1 RM for Leg Extensors | 3 Months
  Changes from the baseline, 1 RM Is used to assess maximum muscle strength. Patient will be asked to perform leg press that is to extend knee against maximum resistance once. weight will be recorded in Kgs.
1 RM for Leg Extensors | 6 Months
  Changes from 3 Months, 1 RM Is used to assess maximum muscle strength. Patient will be asked to perform leg press that is to extend knee against maximum resistance once. weight will be recorded in Kgs.
1 RM for Trunk Extensors | 3 Months
  Changes Baseline, 1 RM Is used to assess maximum muscle strength. Patient will be asked to perform deadlift, maximum weight lifted will be recorded in Kgs.
1 RM for Trunk Extensors | 6 Months
  Changes from 3 Months, 1 RM Is used to assess maximum muscle strength. Patient will be asked to perform deadlift, maximum weight lifted will be recorded in Kgs.
30-second sit to stand test (Reps) | 3 Months
  Changes from Baseline, It involves counting the number of times the participant can rise to a full standing position from the seated position on a chair without using the arms
30-second sit to stand test (Reps) | 6 Months
  Changes from 3 Months, It involves counting the number of times the participant can rise to a full standing position from the seated position on a chair without using the arms
Time up and Go test | 3 Months
  Changes from Baseline, participants will be instructed to walk at usual speed for three meter and then walk back to sit down .Note time on stopwatch .The average of tests trail will be measured as the mean of TUG.
Time up and Go test | 6 Months
  Changes from 3 Months, participants will be instructed to walk at usual speed for three meter and then walk back to sit down .Note time on stopwatch .The average of tests trail will be measured as the mean of TUG.
Dynamic Gait Index | 3 Months
  Changes from Baseline, DGI was Developed to assess the likelihood of falling in older adults. Designed to test eight facets of gait. A four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function. Total Score is 24
Dynamic Gait Index | 6 Months
  Changes from 3 months, DGI was Developed to assess the likelihood of falling in older adults. Designed to test eight facets of gait. A four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function. Total Score is 24
Falls Efficacy Scale | 3 Months
  Changes from Baseline, On a scale from 1 to 10, with 1 being very confident and 10 being not confident at all, patient will be asked how confident are you that you do the given activities without falling. A total score of greater than 70 indicates that the person has a fear of falling.
Falls Efficacy Scale | 6 Months
  Changes from 3Months, On a scale from 1 to 10, with 1 being very confident and 10 being not confident at all, patient will be asked how confident are you that you do the given activities without falling. A total score of greater than 70 indicates that the person has a fear of falling.
Berg balance scale | 3 Months
  Changes from Baseline, The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Berg balance scale | 6 Months
  Changes from 3Months, The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Functional Reach Test (FRT) | 3 Months
  Changes from Baseline, it is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task.In standing, measures the distance between the length of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support.
Functional Reach Test (FRT) | 6 Months
  Changes from 3 months, it is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task.In standing, measures the distance between the length of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, Phd*, Principal Investigator — Riphah International University; Muhammad Naveed Babur, Phd, Study Chair — Isra University islamabad
Locations (2):
- Pakistan (2):
  - Rehab Center RCRAHS Potohar campus, Rawalpindi, Punjab Province
  - Behbud Association of Pakistan, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gianoudis J, Bailey CA, Sanders KM, Nowson CA, Hill K, Ebeling PR, Daly RM. Osteo-cise: strong bones for life: protocol for a community-based randomised controlled trial of a multi-modal exercise and osteoporosis education program for older adults at risk of falls and fractures. BMC Musculoskelet Disord. 2012 May 28;13:78. doi: 10.1186/1471-2474-13-78. PMID 22640372
- [Background] Watson SL, Weeks BK, Weis LJ, Harding AT, Horan SA, Beck BR. High-Intensity Resistance and Impact Training Improves Bone Mineral Density and Physical Function in Postmenopausal Women With Osteopenia and Osteoporosis: The LIFTMOR Randomized Controlled Trial. J Bone Miner Res. 2018 Feb;33(2):211-220. doi: 10.1002/jbmr.3284. Epub 2017 Oct 4. PMID 28975661
- [Background] Watson S, Weeks B, Weis L, Harding A, Horan S, Beck B. High-Intensity Resistance and Impact Training Improves Bone Mineral Density and Physical Function in Postmenopausal Women With Osteopenia and Osteoporosis: The LIFTMOR Randomized Controlled Trial. J Bone Miner Res. 2019 Mar;34(3):572. doi: 10.1002/jbmr.3659. Epub 2019 Feb 25. No abstract available. PMID 30861219
- [Background] Watson SL, Weeks BK, Weis LJ, Horan SA, Beck BR. Heavy resistance training is safe and improves bone, function, and stature in postmenopausal women with low to very low bone mass: novel early findings from the LIFTMOR trial. Osteoporos Int. 2015 Dec;26(12):2889-94. doi: 10.1007/s00198-015-3263-2. Epub 2015 Aug 5. PMID 26243363
- [Background] Watson SL, Weeks BK, Weis LJ, Harding AT, Horan SA, Beck BR. High-intensity exercise did not cause vertebral fractures and improves thoracic kyphosis in postmenopausal women with low to very low bone mass: the LIFTMOR trial. Osteoporos Int. 2019 May;30(5):957-964. doi: 10.1007/s00198-018-04829-z. Epub 2019 Jan 5. PMID 30612163
- [Background] Marques EA, Mota J, Machado L, Sousa F, Coelho M, Moreira P, Carvalho J. Multicomponent training program with weight-bearing exercises elicits favorable bone density, muscle strength, and balance adaptations in older women. Calcif Tissue Int. 2011 Feb;88(2):117-29. doi: 10.1007/s00223-010-9437-1. Epub 2010 Nov 27. PMID 21113584
- [Derived] Riaz H, Babur MN, Farooq A. Effects of high-intensity multi-modal exercise training (HIT-MMEX) on bone mineral density and muscle performance in postmenopausal women. A Pilot randomized controlled trial. J Pak Med Assoc. 2022 Oct;72(10):1904-1908. doi: 10.47391/JPMA.5394. PMID 36660974